CLINICAL TRIAL: NCT05565729
Title: A Phase 1, Randomized, Placebo-controlled, Participant- and Investigator-blind, Single-dose Study of the Pharmacokinetics of LY3471851 Following Subcutaneous Dosing of LY3471851 in Healthy Participants
Brief Title: A Phase I Study of LY3471851 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nektar Therapeutics (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 17603; J1P-MC-KFAN (Other: Eli Lilly and Company)
Record Dates: First submitted 2022-10-03; First posted 2022-10-04 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11-02

CONDITIONS: Healthy
Keywords: Interleukin-2; NKTR-358; Pharmacokinetics
MeSH Terms: interventions — levocetirizine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- LY3471851 (Test formulation) (Experimental): LY3471851 administered subcutaneously (SC).
  Interventions: Drug: LY3471851
- LY3471851 (Test) + Levocetirizine (Experimental): LY3471851 administered SC in combination with levocetirizine given orally.
  Interventions: Drug: LY3471851; Drug: Levocetirizine
- LY3471851 (Reference formulation) (Active Comparator): LY3471851 administered SC.
  Interventions: Drug: LY3471851
- Placebo (Placebo Comparator): Placebo administered SC.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3471851 — Administered SC.
  Other Names: NKTR-358
  Arms: LY3471851 (Reference formulation); LY3471851 (Test formulation); LY3471851 (Test) + Levocetirizine
Drug: Placebo — Administered SC.
  Arms: Placebo
Drug: Levocetirizine — Administered orally.
  Arms: LY3471851 (Test) + Levocetirizine

SUMMARY:
The purpose of this study is to compare two different formulations (test & reference) of LY3471851 in healthy participants. This study will compare how much of each formulation gets into the blood stream and how long it takes the body to remove it. Information about any side effects that may occur will also be collected. Participants will remain in the study for about 12 weeks, after receiving the study drug that is LY3471851.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are overtly healthy as determined by medical history and physical examination
* Have body weight greater than 45 kilograms (kg) and body mass index within the range 18.0 to 32.0 kilograms per square meter (kg/m²)
* Male and female participants must agree to adhere to contraceptive requirements

Exclusion Criteria:

* Have an abnormality in the 12-lead electrocardiogram (ECG), vital signs, or both
* Have had symptomatic herpes zoster within 3 months prior to screening
* Have a known allergy or hypersensitivity to levocetirizine
* Intend to use prescription or nonprescription medication within 14 days or 5 half-lives prior to dosing
* Have received treatment with biologic agents within 3 months or 5 half-lives prior to dosing
* Smoke more than 10 cigarettes or other tobacco products per day before study entry
* Are pregnant or breastfeeding, or intend to become pregnant or breastfeed during the study

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2022-10-05 (Actual); Primary Completion 2023-02-23 (Actual); Study Completion 2023-02-23 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Maximum Concentration (Cmax) of LY3471851 | Predose up to 56 days postdose
  PK: Cmax of LY3471851
PK: Area Under the Concentration Versus Time Curve (AUC) of LY3471851 | Predose up to 56 days postdose
  PK: AUC of LY3471851

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Nektar Therapeutics
Locations (1):
- Covance Dallas, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No